CLINICAL TRIAL: NCT05384197
Title: Enhanced Versus Extended Preoperative Antibiotic Prophylaxis Regimens for Retrograde Intrarenal Surgery in High Infectious Risk Patients: Randomized Controlled Trial
Brief Title: Enhanced Versus Extended Preoperative Antibiotic Prophylaxis Regimens for Retrograde Intrarenal Surgery in High Infectious Risk Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AS-5-2022
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Renal Stone
Keywords: Renal stone; Retrograde intrarenal surgery; Infectious complications; Sepsis
MeSH Terms: conditions — Nephrolithiasis; Sepsis

STUDY DESIGN:
Intervention Model Description: In the available literature, we lack the risk categorization of infectious complications after RIRS with subsequent recommendation as regard to AP in different risk patients. Therefore we are planning to investigate the optimal protocol for AP prior to RIRS in high-risk population through comparing the enhanced regimen (2days) vs. the extended regimen (7 days) in a randomized controlled trial (RCT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced regimen (Active Comparator): They will receive two days antibiotic prophylaxis according to the predetermined protocol.
  Sulfamethoxazole-Trimethoprim (TMP-SMX) twice daily will be utilized as the first choice AP for 2 days according to the assigned randomization group with the last day of AP course being one day prior to intervention.
  In patients with allergy or resistance to TMP-SMX, the following antibiotics will be considered in the following order: 100 mg Nitrofurantoin twice daily, 500 mg Ciprofloxacin twice daily or 200 mg Cefpodoxime twice daily.
  Patients with positive culture which is sensitive only to parenteral antibiotics will receive culture-based intramuscular/intravenous antibiotics following the same schedule (2 days with the last day of AP course being one day prior to intervention)
  Interventions: Drug: Enhanced regimen
- Extended regimen (Active Comparator): They will receive seven days antibiotic prophylaxis according to the predetermined protocol.
  Sulfamethoxazole-Trimethoprim (TMP-SMX) twice daily will be utilized as the first choice AP for 7 days with the last day of AP course being one day prior to intervention.
  In patients with allergy or resistance to TMP-SMX, the following antibiotics will be considered in the following order: 100 mg Nitrofurantoin twice daily, 500 mg Ciprofloxacin twice daily or 200 mg Cefpodoxime twice daily.
  Patients with positive culture which is sensitive only to parenteral antibiotics will receive culture-based intramuscular/intravenous antibiotics following the same schedule ( 7 days with the last day of AP course being one day prior to intervention)
  Interventions: Drug: Extended regimen

INTERVENTIONS:
Drug: Enhanced regimen — Sulfamethoxazole-Trimethoprim (TMP-SMX) twice daily will be utilized as the first choice AP for 2 days with the last day of AP course being one day prior to intervention.
  In patients with allergy or resistance to TMP-SMX, the following antibiotics will be considered in the following order: 100 mg Nitrofurantoin twice daily, 500 mg Ciprofloxacin twice daily or 200 mg Cefpodoxime twice daily.
  Patients with positive culture which is sensitive only to parenteral antibiotics will receive culture-based intramuscular/intravenous antibiotics following the same schedule (2 days with the last day of AP course being one day prior to intervention)
  Arms: Enhanced regimen
Drug: Extended regimen — Sulfamethoxazole-Trimethoprim (TMP-SMX) twice daily will be utilized as the first choice AP for 7 days with the last day of AP course being one day prior to intervention.
  In patients with allergy or resistance to TMP-SMX, the following antibiotics will be considered in the following order: 100 mg Nitrofurantoin twice daily, 500 mg Ciprofloxacin twice daily or 200 mg Cefpodoxime twice daily.
  Patients with positive culture which is sensitive only to parenteral antibiotics will receive culture-based intramuscular/intravenous antibiotics following the same schedule (7 days with the last day of AP course being one day prior to intervention)
  Arms: Extended regimen

SUMMARY:
In the available literature, there is a lack the risk categorization of infectious complications after RIRS with subsequent recommendation as regard to AP in different risk patients. Therefore this study is planning to investigate the optimal protocol for AP prior to RIRS in high-risk population through comparing the enhanced regimen (2days) vs. the extended regimen (7 days) in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Retrograde intrarenal surgery (RIRS) has gained a wide popularity in the management of renal stones due to tremendous technological advancements over the last years. According to the current guidelines, RIRS could be offered as a first line surgical treatment option for renal stones less than 20 mm (or ≤ 10 mm for lower pole stone/s) with favorable stone free rate (SFR).

Despite being a minimally invasive, several morbid complications could be encountered during/after RIRS. Post-operative infectious complications constitute one of the major reported complications after RIRS with varying presentations which include urosepsis, febrile urinary tract infection (UTI) and asymptomatic bacteriuria.

Several large-populations studies have reported the incidence of infectious complications post-RIRS. Among ≈ 12.000 patients undergoing ureteroscopy and were evaluated by The Clinical Research Office of Endourological Society (CROES), post-operative fever, UTI and urosepsis were reported in 1.8%, 1.3% and 0.3%, respectively. Moreover, in another report by Reducing Operative Complications from Kidney stones (ROCK) for 1.817 patients undergoing RIRS, 2.4% required hospital readmission (HR) for infectious complications.

The underlying mechanisms of infectious complications post-RIRS include combination of existing bacteria in the urinary tract and rising intrarenal pressure due to prolonged and/or vigorous irrigation. In addition, several studies have investigated the independent predictors of infectious complications after RIRS with identified positive preoperative urine culture or prior history of recurrent UTI, long-lasting indwelling ureteral stents, diabetes mellitus (DM) and immunocompromised patients.

In addition to the substantial patient morbidity, post-operative infectious complications constitute a major burden to the health care resources. Therefore, minimizing these devastating events should an important consideration by health care providers not only for improving the patient satisfaction but also for cost-saving issues. Therefore, it is a crucial entity for clinicians to identify high-risk patients for post-RIRS infectious complications and to exhaust the different clinical mitigations to minimize these events.

According to American Urological Association (AUA) Best Practice Statements on Antibiotic Prophylaxis (AP), single dose of perioperative antibiotics is indicated for all cases prior to RIRS. However, the exact regimen and duration of preoperative AP for high risk patients for infectious complication are still undefined.

In previous studies on AP for high risk patients prior to percutaneous nephrolithotomy (PCNL), different protocols were compared as regard to its impact on infectious events after PCNL. Despite the reported advantage of the extended regimen on minimizing the infectious events, the drawbacks of prolonged antibiotics as untoward adverse events (AEs) and drug resistance should be considered.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Age ≥18 years.
* Renal stone <20 mm in which RIRS is recommended.
* High susceptibility of post-procedural infectious complications by one or more of the followings: - Positive preoperative urine culture within 12 weeks of the planned intervention. -Indwelling ureteral stents for more than 4 weeks. -Diabetes mellitus.

Exclusion Criteria:

* Solitary kidney.
* Chronic kidney disease.
* Pregnant.
* Have received antibiotics within 7 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative sepsis | 30 days after intervention
  Postoperative sepsis is defined as severe post-procedural (within 12 hours after the procedure with coexisting positive urine culture) infectious complication with ≥ two of the following findings: - Body temperature more than 38.3C or below 36C. - Tachycardia (>90/minute). - Respiratory rate more than 20/minute. - Disturbed mental status. - Systolic blood pressure < 90 mmHg & mean arterial pressure < 70 mmHg or systolic blood pressure decrease < 40 mmHg. - WBC >12,000 or <4,000.

SECONDARY OUTCOMES:
Rate of postoperative fever | 30 days after intervention
Rate of postoperative UTI | 30 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Study Director — Mansoura University; Ehab Nour, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsawy AA, Nour EA, Nabeeh A, El-Nahas AR. Enhanced versus extended preoperative antibiotic prophylaxis for retrograde intrarenal surgery in high infectious risk patients: a randomized controlled trial. World J Urol. 2025 Dec 29;44(1):70. doi: 10.1007/s00345-025-06150-x. PMID 41460253